CLINICAL TRIAL: NCT00250341
Title: Non-Invasive Measures of Distal Lung Disease in Asthmatics Before and After Therapy Directed at the Proximal vs. Distal Lung
Brief Title: Non-invasive Measures of Distal Lung Disease in Asthmatics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IXR-403-4-196
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advair (Active Comparator)
  Interventions: Drug: Advair
- QVAR (Experimental)
  Interventions: Drug: QVAR; Drug: Servent Diskus

INTERVENTIONS:
Drug: QVAR — 480 mcg
  Other Names: beclomethasone dipropionate HFA
  Arms: QVAR
Drug: Advair — 250/50 mcg
  Other Names: Advair Diskus
  Arms: Advair
Drug: Servent Diskus — 50 mcg
  Arms: QVAR

SUMMARY:
This is a Phase 4, single center study conducted in mild-to moderate asthmatics.

DETAILED DESCRIPTION:
The study consists of 3 phases. There are 7 study visits.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Currently using SABA prn or a low-to-moderate persistent asthma

Exclusion Criteria:

* Tobacco use within 1 year or >= 5 pack years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2005-09-30 (Actual); Primary Completion 2007-09-30 (Actual); Study Completion 2007-09-30 (Actual)

PRIMARY OUTCOMES:
High resolution Cat Scans

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Zeidler, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States